CLINICAL TRIAL: NCT07156630
Title: Quick Measure Study for iCare ST500 and iCare IC200
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icare Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TA04-310
Record Dates: First submitted 2025-08-21; First posted 2025-09-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- iCare ST500 and iCare IC200 vs GAT and Tonovera (Experimental)
  Interventions: Device: iCare ST500; Device: iCare IC200; Device: GAT; Device: Tonovera

INTERVENTIONS:
Device: iCare ST500 — Measurement of IOP
Device: iCare IC200 — Measurement of IOP
Device: GAT — Measurement of IOP
Device: Tonovera — Measurement of IOP

SUMMARY:
The aim of this clinical study is to compare the agreement and precision of the intraocular pressure (IOP) results measured with the Quick Measure feature of iCare ST500 and iCare IC200 tonometers with results obtained with reference tonometers (Goldmann applanation tonometry and Tono-Vera tonometer). The data will be collected and evaluated in accordance with ISO 8612:2009 "Ophthalmic Instruments - Tonometers" (at least 120 eyes divided in three IOP groups with a minimum of 40 eyes per group, 95% of the paired differences between the reference tonometer and the test tonometer must fall within the tolerance of ±5 mmHg).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years

Exclusion Criteria:

1. Subjects with only one functional eye
2. Subjects having poor or eccentric fixation in the study eye
3. High corneal astigmatism >3D in the study eye
4. Central corneal scarring
5. History of prior incisional glaucoma surgery or corneal surgery, including corneal refractive laser surgery in the study eye
6. Microphthalmos
7. Buphthalmos
8. Contact lens use within one week of continuous wear and within one hour if lens is worn occasionally
9. Dry eyes (clinically significant)
10. Lid squeezers - blepharospasm
11. Nystagmus
12. Keratoconus
13. Any other corneal or conjunctival pathology or infection relevant to this study
14. Central corneal thickness greater than 600 μm or less than 500 μm in the study eye
15. Cataract Extraction within last 2 months in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2025-08-28 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Demonstrate compliance with ISO 8612:2009-Ophthalmics-Ophthalmic Instruments-Tonometers | Through study completion, estimated 4 months
  Subjects will be distributed into Low IOP, Medium IOP, and High IOP groups based on Goldmann Applanation Tonometer measurements. The iCare ST500 Tonometer and iCare IC200 Tonometer measurements will be within +/-5.0 mmHg of the Goldmann Applanation Tonometer measurements in all groups.

CONTACTS AND LOCATIONS:
Locations (1):
- NVision Clinical Research LLC, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No